CLINICAL TRIAL: NCT05882084
Title: Double Blind Placebo Controlled Oral Supplementation of Astaxanthin on Skin Photoaging, Hydration and Elasticity
Brief Title: Oral Supplementation of Astaxanthin on Skin Photoaging, Hydration and Elasticity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Integrative Skin Science and Research (Industry)
Collaborators: AstaReal (Unknown)
Responsible Party: Principal Investigator, Raja Sivamani, MD MS AP, Principal Investigator, Integrative Skin Science and Research
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Asta_Skin_01
Record Dates: First submitted 2023-05-21; First posted 2023-05-31 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Photoaging
Keywords: Carotenoid; Astaxanthin; Skin; Hydration; Elasticity
MeSH Terms: interventions — astaxanthine

STUDY DESIGN:
Intervention Model Description: Astaxanthin vs Placebo
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Astaxanthin (Experimental): 6 mg daily
  Interventions: Dietary Supplement: Astaxanthin 6 mg daily
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Astaxanthin 6 mg daily — Astaxanthin at 6 mg is given for daily ingestion and compared against placebo.
  Arms: Astaxanthin
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study is a double-blind placebo controlled study to assess whether oral astaxanthin can improve skin hydration, skin elasticity, improve skin pigmentation, and reduce facial redness.

ELIGIBILITY:
Inclusion criteria:

* Females who are 30 to 55 years of age
* Half of the women will have Fitzpatrick skin type 1-3 and the other half of the women will have Fitzpatrick skin type 4-6

Exclusion criteria:

* Individuals with a known allergy to astaxanthin or other carotenoids (such as zeaxanthin, lutein, lycopene).
* Individuals who are unwilling to discontinue carotenoid supplementation for at least 1 month prior to enrollment
* Individuals unwilling to restrict intake of foods like shrimp, salmon, mangos, carrots, and tomatoes during the study.
* New supplementation within 4 weeks with tocopherol
* Individuals who are unwilling to stay consistent with a facial cleansing regimen.
* Those who are unwilling to discontinue topical hydroquinone, retinoid or benzoyl peroxide for 2 weeks prior to enrollment
* Individuals who are pregnant or breastfeeding.
* Individuals who have changed any of their hormonal based contraception within 3 months prior to joining the study.
* Current tobacco smoker or a tobacco smoking history of greater than 10 pack-years

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-07-24 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Skin Hydration | 8 weeks
  Skin hydration measured with a non-invasive device, SkinMoistureMeterSC
Skin elasticity | 8 weeks
  Skin elasticity measured with a non-invasive device, Skin Elastimeter

SECONDARY OUTCOMES:
Facial pigmentation | 8 weeks
  Facial pigment as measured by BTBP facial imaging analysis
Facial redness | 8 weeks
  Facial pigment as measured by BTBP facial imaging analysis

CONTACTS AND LOCATIONS:
Overall Officials: Raja Sivamani, MD, Principal Investigator — Integrative Skin Science and Research
Locations (1):
- Integrative Skin Science and Research, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No